CLINICAL TRIAL: NCT07270497
Title: The Effect of Pharmacotherapy With GLP-1 and GIP/GLP-1 Analogs on Changes in Qualitative and Quantitative Parameters of the Diet as Well as Metabolic and Behavioral Parameters in Patients With Excess Body Weight
Status: Recruiting | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Other Study IDs: KB/136/2025
Record Dates: First submitted 2025-11-14; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: GLP-1; Nutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to comprehensively assess the early and long-term effects of GLP-1 and GIP/GLP-1 analogue medications on metabolic and behavioral parameters, with particular emphasis on qualitative and quantitative dietary changes in patients undergoing treatment for overweight and obesity. Participation in the study will involve four follow-up visits per year at the Clinic of Diabetology and Internal Medicine, Central Clinical Hospital, University Clinical Clinical Hospital, Medical University of Warsaw: before treatment initiation and after 3, 6, and 12 months. The analysis will focus not only on metabolic effects (weight loss, changes in body composition, and improved biochemical parameters), but also on nutritional and behavioral aspects, including diet, appetite regulation, risk of malnutrition and muscle loss, and the occurrence of adverse events. The study will allow for a multifaceted assessment of the impact of treatment with GLP-1 and GIP/GLP-1 analogues on patients with excess body weight.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years,
* Diagnosed obesity (BMI ≥ 30 kg/m²) or overweight (BMI ≥ 27 kg/m²) with comorbidities associated with excess body weight (including type 2 diabetes, hypertension, dyslipidemia, obstructive sleep apnea, cardiovascular disease),
* Eligibility for treatment with GLP-1 or GIP/GLP-1 analogues,
* Not taking GLP-1 and GIP/GLP-1 analogue medications for at least one year prior to study enrollment,
* Ability to provide informed consent,
* Informed consent to participate in the study.

Exclusion Criteria:

* Age under 18 or over 65 years,
* Inability to qualify for treatment with GLP-1 and GIP/GLP-1 analogues,
* Pregnancy or breastfeeding,
* Diagnosed eating disorders,
* Active cancer or gastrointestinal conditions that may affect the absorption or tolerance of treatment (e.g., inflammatory bowel disease, conditions after extensive gastrointestinal resections, conditions after bariatric surgery),
* Inability to participate in regular follow-up visits,
* Inability to provide informed consent,
* Failure to provide informed consent to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People diagnosed with obesity (BMI ≥ 30 kg/m²) or overweight (BMI ≥ 27 kg/m²) with comorbidities associated with excess body weight (including type 2 diabetes, hypertension, dyslipidemia, obstructive sleep apnea, cardiovascular disease), eligibilited for treatment with GLP-1 or GIP/GLP-1 analogues.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-08-14 (Estimated); Study Completion 2026-08-14 (Estimated)

PRIMARY OUTCOMES:
change in body weight | 12 months
  percentage change in body weight from baseline to the end of follow-up

SECONDARY OUTCOMES:
Change in lean body mass | 12 months
  Change in lean body mass measured using the Tanita MC-980MA Plus segmental body composition analyzer. Reported in kilograms (kg).
Change in total fat mass | 12 months
  Change in total fat mass measured using the Tanita MC-980MA Plus segmental body composition analyzer (bioelectrical impedance analysis). Reported in kilograms (kg).
Change in percent body fat | 12 months
  Change in percent body fat measured using the Tanita MC-980MA Plus segmental body composition analyzer. Reported as percent of total body mass (%).
Change in HbA1c | 12 months
  Change in hemoglobin A1c measured in venous blood using standard laboratory HPLC assay. Reported as percent (%).
Change in fasting plasma glucose | 12 months
  Change in fasting plasma glucose measured using enzymatic laboratory assay. Reported in mmol/L (or mg/dL).
Change in fasting insulin concentration | 12 months
  Change in fasting insulin measured using immunoassay (e.g., ELISA/chemiluminescence). Reported in μU/mL.
Change in HOMA-IR | 12 months
  Change in insulin resistance calculated using HOMA-IR (fasting insulin × fasting glucose / 22.5).
Change in lipid profile | 12 months
  Change in total cholesterol, LDL-C, HDL-C, and triglycerides measured using standard serum laboratory assays. Reported in mmol/L (or mg/dL).
Change in liver enzymes and creatinine | 12 months
  Change in ALT, AST (U/L) and serum creatinine (µmol/L) measured using standard laboratory methods.
Change in daily energy intake | 12 months
  Change in average daily energy intake assessed from 3-day food records (2 weekdays + 1 weekend day), analyzed using a 3-day food diary
Change in diabetes treatment | 12 months
  Number and percentage of participants with changes in diabetes pharmacotherapy (dose modification, medication initiation/discontinuation, or class switch).
Change in antihypertensive treatment | 12 months
  Number and percentage of participants with changes in antihypertensive therapy (dose adjustment, medication initiation/discontinuation, or class switch).
Change in daily carbohydrate intake | 12 months
  Change in daily carbohydrate intake assessed using a 3-day weighed food record and analyzed with validated dietary software. Reported in grams/day and as percent of total energy intake.
Change in daily fat intake | 12 months
  Change in total fat intake assessed using a 3-day weighed food record. Reported in grams/day and percent of total energy intake.
Change in daily protein intake | 12 months
  Change in protein intake assessed using a 3-day weighed food record. Reported in grams/day and grams per kilogram of body weight.
Change in diet quality score (KomPAN) | 12 months
  Change in diet quality assessed using the validated KomPAN questionnaire (modified for 3-month frequency assessment). Reported as the KomPAN dietary index score, according to validated scoring rules.
Change in frequency of consumption of selected food groups | 12 months
  Change in the frequency of consumption of selected food groups assessed using the validated KomPAN food frequency questionnaire. Includes changes in consumption of: vegetables, fruit, whole grains, sweets, high-fat foods, meat products, sweetened beverages, and others defined in KomPAN. Reported as frequency categories or converted frequency units.
Change in emotional eating score (TFEQ-R18) | 12 months
  Change in emotional eating assessed with the validated Three-Factor Eating Questionnaire (TFEQ-R18). Scale range 0-100 (converted), higher scores indicate stronger emotional eating tendencies.
Change in uncontrolled eating score (TFEQ-R18) | 12 months
  Change in uncontrolled eating assessed using TFEQ-R18. Higher scores indicate greater susceptibility to uncontrolled eating.
Change in cognitive restraint score (TFEQ-R18) | 12 months
  Change in cognitive restraint (intentional food restriction) assessed using TFEQ-R18. Higher scores indicate higher restraint.
Change in subjective hunger (VAS) | 12 months
  Change in subjective hunger measured using a Visual Analog Scale (VAS, 0-100 mm) within the validated questionnaire set. Higher scores indicate greater hunger
Change in subjective satiety (VAS) | 12 months
  Change in subjective satiety measured using VAS (0-100 mm). Higher scores indicate greater satiety.
Change in sweet taste preference (VAS) | 12 months
  Change in desire to consume sweet foods measured using a Visual Analog Scale (VAS, 0-100 mm) as part of the custom taste preference questionnaire.
Change in preference for high-fat foods (VAS) | 12 months
  Change in desire to consume high-fat foods measured using VAS (0-100 mm).
Change in preference for salty foods (VAS) | 12 months
  Change in desire to consume salty foods measured using VAS (0-100 mm).
Change in preference for meat-based products (VAS) | 12 months
  Change in desire to consume meat-based foods measured using VAS (0-100 mm).
Change in preference for fresh/fruit-based foods (VAS) | 12 months
  Change in desire to consume fresh or fruit-based foods assessed using VAS (0-100 mm).
Change in risk of inadequate nutrient intake | 12 months
  Change in risk of insufficient intake of key nutrients (vitamin D, B12, folate, iron, protein) assessed indirectly through 3-day weighed food records and KomPAN questionnaire data. Reported as intake relative to recommended dietary allowances.
Change in meal frequency | 12 months
  Change in number of daily eating occasions based on the 3-day food record. Reported as meals/day.
Change in mean daily step count | 12 months
  Change in average daily number of steps recorded from the participant's smartphone health application. Step count is extracted from the app's built-in accelerometer-based activity tracking. Reported as steps per day.
Change in handgrip strength | 12 months
  Change in maximal handgrip strength measured using a calibrated handheld dynamometer. Strength is assessed in the dominant hand, with three attempts per measurement, and the highest value recorded. Reported in kilograms (kg).

CONTACTS AND LOCATIONS:
Locations (1):
- Klinika Diabetologii i Chorób Wewnętrznych Uniwersyteckiego Centrum Klinicznego Warszawskiego Uniwersytetu Medycznego, Warsaw, Warszawa, Poland